CLINICAL TRIAL: NCT01244789
Title: A Phase II Randomized Trial of Postoperative Chemotherapy or no Further Treatment for Patients With Node-negative Stage I-II Intermediate or High Risk Endometrial Cancer
Brief Title: Chemotherapy or Observation in Stage I-II Intermediate or High Risk Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Danish Gynecological Cancer Group (Network)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Arbeitsgemeinschaft Gynaekologische Onkologie Austria (Other); North Eastern German Society of Gynaecological Oncology (Other); Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other); Belgian Gynaecological Oncology Group (Other); Mario Negri Gynecologic Oncology group (MaNGO) (Other); Israeli Society of Gynecologic Oncology (Other); Multicenter Italian Trials in Ovarian cancer and gynecologic malignancies (MITO) (Unknown); Central and Eastern European Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-EN2-DGCG; 2010-023081-52 (EudraCT Number)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; chemotherapy; carboplatin; paclitaxel; Stage 1 & 2; node-negative; intermediate risk; high risk
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (Active Comparator): postoperative observation only
  Interventions: Other: observation
- Combination chemotherapy (Experimental): postoperative 6 courses of 3 weekly iv carboplatin-paclitaxel combination chemotherapy
  Interventions: Drug: carboplatin and paclitaxel

INTERVENTIONS:
Drug: carboplatin and paclitaxel — 6 courses of iv 3-weekly chemotherapy Carboplatin AUC5 Paclitaxel 175mg/m2
  Arms: Combination chemotherapy
Other: observation — active observation
  Arms: Observation

SUMMARY:
Patients with stage 1 & 2 endometrial cancer are treated with surgery. Despite the fact that disease is confound to uterus, unfortunately some of these patients may relapse and die of their disease. Postoperative radiotherapy cannot improve survival. Chemotherapy has shown survival benefit in more advanced stage disease (stage 3 & 4).

This study evaluates if one can improve survival in intermediate and high risk early-stage patients by offering them postoperative chemotherapy. This is a randomized phase 3 trial where effect of postoperative chemotherapy is compared with postoperative observation alone (standard strategy).

Substudy: Translational research

DETAILED DESCRIPTION:
Patients with medium and high risk stage I and II endometrial cancers have, despite radical surgery, a rather high risk for progression.

Adjuvant radiotherapy was the traditional therapy for many decades. Four randomized phase III studies and a meta-analysis have revealed that adjuvant radiotherapy improves local control at the cost of excessive short and long term toxicity, though has absolutely no impact on survival.

Two phase III studies have randomized between adjuvant radiotherapy versus adjuvant chemotherapy, both failed to show any difference in survival between radiotherapy and chemotherapy, though both studies are criticized for inferior chemotherapy regimens or inclusion of good prognosis patients. The GOG-122 study on more advanced cases (stage 3 & 4) randomized between combination chemotherapy versus whole abdominal irradiation and found significant improvement in survival in the chemotherapy arm.

NSGO-EC-9501 and MaNGO studies have indicated that adjuvant chemotherapy added to adjuvant radiotherapy may improve survival compared to adjuvant radiotherapy alone in early stage medium and high risk patients. One may conclude that impact on survival comes only from chemotherapy. Many investigators have therefore adapted adjuvant chemotherapy as standard treatment in various countries including Denmark. However, such conclusion has low level of evidence, as there are no randomized phase III studies comparing postoperative observation alone versus adjuvant chemotherapy.

It is of utmost importance to demonstrate efficacy of adjuvant combination chemotherapy in a randomized phase III trial comparing to no further treatment in the medium and high risk node negative stage 1 & 2 patients.

Combination chemotherapy regimen of paclitaxel-carboplatin is proposed in this study, as this combination is effective and well tolerated.

The eligible patients for such a study are a fraction of patients with endometrial cancer therefore this study will be performed within the ENGOT collaboration.

ELIGIBILITY:
Inclusion Criteria:

Target Population

1. Only node-negative patients are eligible: Histological confirmed endometrial carcinoma with no macroscopic remaining tumour after primary surgery and lymph-node negative disease, with one of the following postoperative FIGO 2009 stage and grade:

   1. Stage I grade 3 endometrioid adenocarcinoma
   2. Stage II endometrioid adenocarcinoma
   3. Stage I and II type 2 histology (clear cell, serous, squamous cell carcinoma, or undifferentiated carcinoma) Prior therapy
2. Patients have undergone hysterectomy (total abdominal hysterectomy, radical hysterectomy, laparoscopic or robotic hysterectomy) and bilateral salpingo-oophorectomy (BSO) and pelvic lymphadenectomy (LNE).
3. LNE: minimum 12 pelvic nodes (6 from each side) should be removed. Para-aortic LNE is optional
4. Omentectomy strongly recommended in clear cell, serous or undifferentiated carcinoma.
5. Surgery performed within 10 weeks of randomization. If the dates for hysterectomy and lymph node dissection are different, 10 weeks are counted from the last surgery, and in that case the gap between two surgeries should not exceed 8 weeks.

   Other inclusion criteria
6. Patients must give informed consent according to the rules and regulations of the individual participating centres
7. Patients have not received any other anticancer therapy other than surgery.
8. Adjuvant vaginal brachytherapy is permitted in both arms. In chemotherapy arm, timing of VBT should not cause delay in chemotherapy delivery.
9. Patients must have a WHO performance status of 0-2
10. Patients must have an adequate bone-marrow, renal and hepatic function (WBC ≥3.0x109/L, neutrophils ≥1.5x109/L, platelets ≥100x109/L, total S-bilirubin <2 x upper normal value, ALAT <2.5 x upper normal value, estimated GFR >50 ml/min (measured or calculated according to Cockroft-Gault or Jeliffe). Up to 5% deviation for hematological values and 10% deviation for s-bilirubin and ALAT are tolerated.
11. Life expectancy of at least 12 weeks
12. Patients must be fit to receive combination chemotherapy
13. Patient's age >18 years

Exclusion criteria:

Target Disease Exceptions

1. Carcinosarcoma, Sarcomas or small cell carcinoma with neuroendocrine differentiation.

   Prohibited Treatments and/or Therapies
2. External Beam Radiotherapy
3. Concurrent cancer therapy
4. Concurrent treatment with an anticancer investigational agent or participation in another anticancer clinical trial Other exclusion criteria
5. Previous or concurrent malignant disease except for curatively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin
6. Active infection or other serious underlying medical condition, which might prevent the patient from receiving treatment or to be followed
7. Whatever reasons which interferes with an adequate follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | May 2017
  To detect an overall absolute difference in five-year survival of 10%, from 72% to 82%, at the 2.5% level with 80% power, 135 deaths corresponding to 644 patients are needed. Assuming a dropout rate of 5%, 678 patients have to be accrued, leaving 644 patients for the overall analysis.

SECONDARY OUTCOMES:
Overall Survival in endometrioid subgroup | May 2017
  In the endometrioid subgroup an absolute difference in five-year survival of 12%, from 74% to 86% is expected. Assuming this, 79 deaths corresponding to 438 patients are needed to yield 80% power at the 2.5% level. Assuming a dropout rate of 5%, 678 patients have to be accrued, leaving 644 patients for the overall analysis and 75% of these, or 483 patients, for the analysis in the endometrioid subgroup.
Disease Specific Survival | May 2017
  Exploratory endpoint
Progression-Free Survival | May 2017
  Exploratory endpoint
Toxicity - Acute toxicity (0-6 months from randomization). Late toxicity is registered during whole study period. | May 2017
  Acute toxicity (0-6 months from randomization). Late toxicity is registered during whole study period. Exploratory endpoint
QOL, EORTC QLQ-30 | May 2017
  EORTC QLQ-30
EORTC QLQ-EN-24 | may 2017
  QLQ EORTC QLQ-EN-24
Rate of isolated pelvic relapse | May 2017
  Exploratory endpoint
Rate of isolated distant relapse | May 2017
  Exploratory endpoint
Rate of mixed (local & distant) relapses | May 2017
  Exploratory endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor R Mirza, MD, Study Chair — Danish Gynecological Cancer Group
Locations (1):
- Danish Gynecological Cancer Group (DGCG), Copenhagen, Denmark